CLINICAL TRIAL: NCT04808830
Title: Prevalence of Musculoskeletal Pain and Its Impact on Quality of Life and Functional Exercise Capacity in Patients With Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Izmir Bakircay University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melih Zeren, Assist. Prof. Dr., Izmir Bakircay University
Other Study IDs: bakircaymzeren02
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary arterial hypertension: Adult patients with pulmonary arterial hypertension
  Interventions: Other: Evaluation of musculoskeletal pain prevalence; Other: Evaluation of quality of life; Other: Evaluation of functional exercise capacity; Other: Evaluation of physical activity level

INTERVENTIONS:
Other: Evaluation of musculoskeletal pain prevalence — Prevalence of musculoskeletal pain will be evaluated over 9 body regions using The Nordic Musculoskeletal Questionnaire.
Other: Evaluation of quality of life — Quality of life will be evaluated using The EmPHasis-10 questionnaire and The Minnesota Living with Heart Failure Questionnaire.
Other: Evaluation of functional exercise capacity — Functional exercise capacity will be evaluated using 6-min walk test.
Other: Evaluation of physical activity level — Physical activity level will be evaluated using International Physical Activity Questionnaire- Short Form

SUMMARY:
Prevalence of musculoskeletal pain and its impact of quality of life and functional exercise capacity will be evaluated in patients with pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Although main symptoms of pulmonary arterial hypertension (PAH) include shortness of breath and exercise intolerance, patients may also experience symptoms related to musculoskeletal system such as muscle fatigue or pain. Due to insufficient cardiac output and chronic arterial hypoxemia, oxygen cannot be delivered to skeletal muscles sufficiently, especially during exertion. In addition, inflammation, which is thought to play an important role in pulmonary vascular remodeling and disease pathophysiology in these patients, affects skeletal muscles as well. Increased sympathetic tone in PAH restricts the perfusion of skeletal muscle by increasing peripheral vascular resistance. With the addition of physical inactivity to all these factors, skeletal muscle metabolism is further impaired. Furthermore, drugs used for the treatment of PAH may induce musculoskeletal pain as a side effect. Musculoskeletal pain is one of the most important factors impairing individual's quality of life, regardless of whether there is an underlying disease. Our aim in this study is to evaluate pain prevalence in the musculoskeletal system over 9 body regions, to compare the pain prevalence of patients using different types of PAH drugs and to examine impact of musculoskeletal pain on quality of life and functional capacity in patients with PAH.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulmonary arterial hypertension

Exclusion Criteria:

* Diagnosis of heart failure or any chronic respiratory disease
* Recent coronary bypass surgery
* Recent acute myocardial infarction
* Having a pacemaker
* Having any orthopedic or neurologic diseases which may impede walking or exercising

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with pulmonary arterial hypertension
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The Nordic Musculoskeletal Questionnaire | At baseline
  The Nordic Musculoskeletal Questionnaire will be used to evaluate musculoskeletal pain prevalence.

SECONDARY OUTCOMES:
The EmPHasis-10 questionnaire | At baseline
  The EmPHasis-10 questionnaire will be used to measure quality of life.
The Minnesota Living with Heart Failure Questionnaire | At baseline
  The Minnesota Living with Heart Failure Questionnaire will be used to measure quality of life.
6-min walk distance | At baseline
  Distance walked in six minutes will be recorded. Test will be conducted according to the guideline of American Thoracic Society (ATS).
International Physical Activity Questionnaire - Short Form | At baseline.
  International Physical Activity Questionnaire - Short Form will be used to measure physical activity level

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Institute of Cardiology, Istanbul, Turkey (Türkiye)